CLINICAL TRIAL: NCT06218810
Title: Cadonilimab in Combination With Bevacizumab and FOLFOX Regimen for the First-Line Treatment of Advanced Unresectable MSS-Type, RAS-Mutated Metastatic Colorectal Cancer: A Single-Arm, Open-Label, Multicenter Phase II Study
Brief Title: Cadonilimab in Combination With Bevacizumab and FOLFOX Regimen for the First-Line Treatment of Advanced Unresectable MSS-Type, RAS-Mutated Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Director, Head of Department of Colorectal Surgery, Principal Investigator, Clinical Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cadolinimab on MSS mCRC
Record Dates: First submitted 2023-12-21; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Colorectal Cancer; Microsatellite Stable Colorectal Carcinoma; RAS Mutation; Cadonilimab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): This study includes only on experimental arm
  Interventions: Drug: Cadonilimab + bevacizumab + FOLFOX

INTERVENTIONS:
Drug: Cadonilimab + bevacizumab + FOLFOX — Cadonilimab + bevacizumab + FOLFOX

SUMMARY:
The dual immunotherapy regimen significantly outperformed previous chemotherapy or immunomonotherapy for MSS type advanced CRC in two key efficacy indicators, ORR and PFS. Researchers have also conducted in-depth analysis of patient transcriptomics, immune microenvironment characteristics, and other related information, which is expected to guide more accurate immune combination therapy for CRC in the future. Our team plans to conduct a multicenter, prospective, single arm clinical trial in patients with RAS mutant MSS unresectable metastatic colorectal cancer, with a focus on observing the 1-year progression free survival rate of the combination of two chemotherapy drugs, bevacizumab and Cadonilimab, as well as ORR, perioperative safety, and long-term survival.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign a written ICF.
2. Age at enrollment: ≥ 18 years old, ≤ 75 years old, both male and female.
3. The Eastern Cancer Collaborative Organization (ECOG) has a physical fitness score of 0 or 1.
4. The expected survival period is ≥ 3 months.
5. Subjects diagnosed with metastatic colorectal adenocarcinoma by histology or cytology.
6. Colorectal cancer patients who have not received systematic anti-tumor therapy in the past and are not suitable for radical surgical resection or local treatment.
7. Genetic testing results indicate pMMR or MSS; RAS mutation;
8. According to RECIST v1.1, there is at least one measurable lesion that is suitable for repeated and accurate measurements. Note: Brain metastases cannot be used as target lesions; For lesions that have received radiation therapy before, it is not recommended to select them as target lesions. If there are no other lesions that meet the target lesion criteria, and the lesion can be measured according to RECIST v1.1 and there is objective evidence to prove significant progression after radiation therapy, the irradiated lesion can be considered as a target lesion.

Exclusion Criteria:

1. Patients with known MSI-H or dMMR.
2. Participants of RAS wild-type.
3. Subjects suffered from other malignant tumors within 3 years before enrollment, except for cured local tumors (such as basal cell skin cancer, squamous cell skin cancer, superficial bladder cancer, cervical carcinoma in situ, etc.).
4. Simultaneously enroll in another clinical study, unless it is an observational, non-interference clinical study or a follow-up period of an intervention study.
5. Received systematic anti-tumor therapy (chemotherapy) within 3 weeks prior to the first administration; Palliative local treatment was performed on non target lesions within 2 weeks prior to the first administration; Received non-specific immunomodulatory therapy (such as interleukin, interferon, thymosin, etc., excluding IL-11 used to treat thrombocytopenia) within 2 weeks before the first administration; Chinese herbal medicine or traditional Chinese patent medicines and simple preparations with anti-tumor indications was received within 1 week before the first administration.
6. Have received any immunotherapy against tumors in the past, including immune checkpoint inhibitors (such as anti-PD-1 antibodies, anti-PD-L1 antibodies, anti-CTLA-4 antibodies, etc.), immune checkpoint agonists (such as ICOS, CD40, CD137, GITR, OX40 antibodies, etc.), immune cell therapy, and any treatment targeting the immune mechanism of tumors.
7. Patients with active autoimmune diseases that require systematic treatment within the past two years (such as using medication to improve the condition, corticosteroids, immunosuppressive agents), and replacement therapy (such as thyroid hormone, insulin, or physiological corticosteroid replacement therapy for adrenal or pituitary dysfunction) are not considered as systematic treatment.
8. A history of active or previous inflammatory bowel disease (such as Crohn's disease, ulcerative colitis, or chronic diarrhea).
9. History of immunodeficiency; HIV antibody test positive individuals; Currently using systemic corticosteroids or other immunosuppressants for a long time.
10. Subjects who are known to have active pulmonary tuberculosis (TB) and suspected to have active TB need to undergo clinical examination to exclude them; Known active syphilis infection.
11. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
12. Previous or current non infectious pneumonia/interstitial lung disease requiring systemic glucocorticoid treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
1-year Progression Free Survival rate | 12 months

SECONDARY OUTCOMES:
AE rate | 24months
  Adverse event incidence rate
ORR | 24months
  Objective response rate
NED | 24months
  No evidence of disease
PFS PFS | 24months
  Progression free survival
OS | 24months
  Overall survival
irORR | 24months
  immune-related objective response rate

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan hosptial, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No